CLINICAL TRIAL: NCT06563973
Title: The Effect of Breast Milk Odor Applied Before First Oral Feeding on Feeding Performance in Preterm Infants
Brief Title: The Effect of Breast Milk Odor on Feeeding in Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Canan Genç, Research Assistant, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2022/0715
Record Dates: First submitted 2024-08-19; First posted 2024-08-21 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Bottle Feeding; Preterm İnfant
Keywords: Feeding Performance; Preterm Infants; Milk Odor
MeSH Terms: conditions — Bottle Feeding; Premature Birth | interventions — Pacifiers

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Breast milk odor and pacifier group (Experimental): A pacifier was given for 3 minutes one hour before feeding and for 2 minutes 10 minutes before feeding to support oral feeding. In contrast to the control group, 2 cc of breast milk was dripped onto a sterile sponge one hour before feeding and placed in the baby's incubator, close to the nose (3 cm away). Heart rate and oxygen saturation levels were recorded 10 minutes before feeding.
  Interventions: Other: Milk odor; Other: Pacifier
- Pacifier group (Active Comparator): A pacifier was provided for 3 minutes one hour before feeding and for 2 minutes 10 minutes before feeding to support oral feeding. Heart rate and oxygen saturation levels were recorded 10 minutes prior to feeding.
  Interventions: Other: Pacifier

INTERVENTIONS:
Other: Milk odor — One hour before feeding time, 2 cc of breast milk was dripped onto a sterile sponge and placed inside the baby's incubator, close to the baby's nose (3 cm).
  Arms: Breast milk odor and pacifier group
Other: Pacifier — To support oral feeding, a pacifier was given for 3 minutes one hour before feeding time and for 2 minutes 10 minutes before feeding time.

SUMMARY:
This study was conducted as a randomized controlled experiment to assess the impact of breast milk odor, applied before the first oral feeding of preterm infants transitioning to oral feeding, on their feeding performance. Infants in the neonatal intensive care unit who were beginning oral feeding were randomly assigned to one of two groups through computer randomization. In the "pacifier" group, infants were given a pacifier for 3 minutes one hour before feeding and again for 2 minutes 10 minutes before feeding to support oral feeding. In contrast, the "breast milk odor and pacifier" group received 2 cc of breast milk, which was dripped onto a sterile sponge and placed about 3 cm from the infant's nose one hour before feeding. At feeding time, all infants in both groups were bottle-fed by the researcher. This marked their first experience with oral feeding. The infants' feeding skills and performance were then evaluated using the Early Feeding Skills (EFS) form during the feeding session.

DETAILED DESCRIPTION:
Detailed Description:

Recent research has indicated that olfactory stimulation can serve as an effective nonpharmacological method for enhancing feeding outcomes. Using breast milk for olfactory stimulation is both a cost-efficient and noninvasive approach that may speed up the process of oral feeding and lead to better feeding results. This study aimed to assess the impact of breast milk odor, applied before the first oral feeding of preterm infants transitioning to oral feeding, on their feeding performance. The sample size was calculated using power analysis, based on data from similar studies. As per the analysis, the study intended to include a total of 50 preterm infants, with at least 25 infants in each group. Following verbal and written consent from the families of eligible infants, the study proceeded with those mothers and infants who agreed to participate.

Before Feeding A pulse oximeter was attached to the feet of all infants to monitor their heart rate and oxygen saturation levels. The researcher filled out the "Preterm Infant Identification Form." Nurses caring for the infants included in the study were briefed, and care was provided for 60 minutes before feeding and 10 minutes after feeding to ensure the babies could rest. No painful or stressful procedures were conducted during this period. All interventions were carried out by the researcher in a quiet and calm environment within the incubator to minimize the impact of external factors. Sixty minutes before feeding, all infants were positioned in a semi-elevated side-lying position.

Pacifier Group: To support oral feeding, a pacifier was provided for 3 minutes one hour before feeding time and again for 2 minutes 10 minutes before feeding. Heart rate and oxygen saturation levels were recorded 10 minutes before feeding.

Breast Milk Scent and Pacifier Group: Similar to the pacifier group, infants in this group received a pacifier for 3 minutes one hour before feeding and for 2 minutes 10 minutes before feeding. Additionally, 2 cc of breast milk was dripped onto a sterile sponge and placed inside the incubator, approximately 3 cm from the infant's nose. Heart rate and oxygen saturation levels were also recorded 10 minutes before feeding.

During Feeding:

Once all pre-feeding procedures were completed and documented, the infant's position remained unchanged by the researcher. The bottle was introduced near the infant's mouth while they were in a semi-raised, side-lying position. The stopwatch was activated as soon as the infant began sucking. To avoid tiring the infant, feeding was limited to 30 minutes. Throughout this period, heart rate (HR) and oxygen saturation (SpO2) were continuously monitored. The infant's feeding skills were assessed using the Early Feeding Skills (EFS) form by an observer nurse who was not involved in the study.

A slow-flow, soft nipple bottle with a smaller hole was used for feeding. To encourage feeding, the researcher gently touched the infant's lips with the bottle nipple. Once the infant's mouth opened, the nipple was placed inside, carefully lowering the tongue. During feeding, any stimulating actions, such as moving or rotating the bottle in the mouth, were avoided.

The infants were closely monitored for signs of fatigue (e.g., reduced sucking, milk leakage, difficulty maintaining posture) and symptoms of physiological or behavioral stress (e.g., pulling the head back, trying to turn away, coughing, grimacing, aspiration, desaturation, apnea, bradycardia, tachycardia). If any stress or fatigue signs were observed, feeding was paused to allow the infant to rest. Feeding resumed once the infant was physiologically stable (HR 120-160/min, SpO2 ≥90) and behaviorally ready.

After Feeding:

To avoid influencing physiological measurements, no interventions were made for 10 minutes post-feeding. The infant's HR, SpO2 values, feeding duration, and the amount of milk consumed during feeding were recorded on the data form.

ELIGIBILITY:
Inclusion Criteria:

parents must give voluntary consent to participate; the infant must have been born between 26 and 34 weeks of gestation, as determined by the mother's last menstrual period; at the time of the study, the infant must be more than 30 weeks postmenstrual; the infant must be transitioning from enteral to oral feeding for the first time; the infant must be free of health issues other than prematurity; the infant must be fed with the mother's milk; the physician must have approved the infant's readiness for oral feeding; the infant must exhibit physiological and behavioral signs that indicate readiness for oral feeding.

Exclusion Criteria:

severe bronchopulmonary dysplasia; any gastrointestinal, neurological, or genetic disorder (such as necrotizing enterocolitis, intracranial hemorrhage, hydrocephalus, omphalocele, Down syndrome, gastroschisis); any condition that could interfere with oral feeding (such as cleft palate, cleft lip, facial muscle paralysis, craniofacial anomaly).

Ages: 26 Weeks to 30 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2023-04-18 (Actual); Primary Completion 2023-11-24 (Actual); Study Completion 2023-11-24 (Actual)

PRIMARY OUTCOMES:
Early Feeding Skills | during feeding up to 1 hour
  An observer nurse, who was not part of the research team, evaluated the infant's feeding skills using the Early Feeding Skills (EFS) Evaluation Form.
The feeding duration (Feeding performance) | immediately after feeding
  The infant's feeding performance was assessed by calculating the feeding duration. To measure feeding time, a stopwatch on a phone was activated at the start of feeding and stopped once feeding concluded.
Feeding performance | immediately after feeding
  The infant's feeding performance was assessed by calculating the amount of food consumed per minute. The total amount of food the infant consumed (in cc) was then compared to the amount prescribed by the doctor.

CONTACTS AND LOCATIONS:
Overall Officials: Duygu Gözen, Prof., Principal Investigator — Koç University
Locations (1):
- Fenerbahce University, Istanbul, İ̇stanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No